CLINICAL TRIAL: NCT05070286
Title: A Lifestyle Weight Management Program for Paediatric Patients With Demyelinating Conditions: Interviews and Stakeholder Meetings.
Brief Title: Lifestyle Weight Management Program: Interviews and Stakeholder Meetings.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oxford Brookes University (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Helen Dawes, Prof Helen Dawes, Oxford Brookes University
Other Study IDs: F.02.2019.13
Record Dates: First submitted 2021-05-11; First posted 2021-10-07 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica
Keywords: Paediatric
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Young people with MS and NMOSD: Young people aged 10-25 years, who were diagnosed with MS or NMOSD prior to the age of 18.
  Semi-structured interviews.
  Interventions: Behavioral: Observational Study.
- Parents of young people with MS and NMOSD: Parents of young people aged 10-25 who were diagnosed with MS or NMOSD prior to the age of 18.
  Semi-Structured Interviews
  Interventions: Behavioral: Observational Study.
- Clinicians: Health care practitioners from medical, nursing and AHP backgrounds with at least two years' experience in NMOSD and MS.
  Interventions: Behavioral: Observational Study.

INTERVENTIONS:
Behavioral: Observational Study. — Semi-structured interviews.

SUMMARY:
Background: An assessment by paediatric neurologists specializing in demyelinating conditions brought attention to the rapid weight change seen among patients recently diagnosed with, and receiving therapy for, neuromyelitis optica spectrum disorder (NMOSD) and multiple sclerosis (MS). An overview of the current literature pinpointed weight change as a concern, and identified fatigue and fear as limiting factors for participation in physical activity, with BMI trajectories in this population significantly higher compared to healthy peers. A look at current patient data highlighted extreme NMOSD cases where some patients' weight doubled in two years. There is currently no available research that addresses weight change and management in paediatric MS or NMOSD patients, but there is research to highlight the importance of maintaining health behaviours. The aim of this research is to co-develop a comprehensive lifestyle weight management program for this cohort.

Methods: Unpinned by the Medical Research Council guidance for developing complex interventions, this research will involve a fourfold approach. It will build on a previously completed systematic review, and a secondary data analysis of current clinical data regarding weight changes in these populations. Semi-structured interviews will be conducted with patients, parents and clinicians in order to obtain qualitative data regarding the collective perspectives of nutrition, weight change and overall health. A list of factors will be identified and presented in a logic model. A program will then be designed, informed by previously gathered information and will be reviewed by a group of stakeholders via stakeholder meetings. This will output a program design, implementation and evaluation plan which will then be evaluated for feasibility. Recruitment, participation, implementation and adherence to the program will be tested. A patient, public involvement (PPI) approach will be taken, with a PPI panel of experts overseeing and guiding the project for its duration.

Results: The results of this research will output a primary version of the lifestyle weight management program for paediatric patients with demyelinating conditions, ready for a feasibility trial.

DETAILED DESCRIPTION:
RESEARCH QUESTIONS AND AIMS

Aim:

To co-develop a comprehensive lifestyle weight management program catered specifically for paediatric patients with demyelinating conditions such as multiple sclerosis (MS) and neuromyelitis optica spectrum disorder (NMOSD).

Objectives:

1. To explore perspectives and perceptions regarding weight change, health and quality of life, through semi-structured interviews of young people with MS and NMOSD, their parents and clinicians.
2. To establish a list of factors that contribute to weight change in the paediatric MS and NMOSD patients following steroid treatment, mapped out in a logic model.
3. To co-design a lifestyle weight management program for paediatric MS and NMOSD patients through the compilation of information and data obtained, and the input from stakeholder meetings.

Outcome:

The final outcome of this study will be a lifestyle weight management program that is ready for a feasibility trial. It will output a set of end-user requirements as well as a fully formed underpinning logic model.

STUDY DESIGN and METHODS of DATA COLLECTION AND DATA ANALYIS

Method overview:

Building on a previously completed scoping review, and an audit of the research team's pre-existing patient data and information from the collaborating institutions, this stage of the research involves three distinct phases:

* Phase 1) Foundational co-development- Interviews
* Phase 2) Logic model of factors
* Phase 3) Program design and implementation plan- Stakeholder Meetings

Phase 1: Interviews. Young people with MS or NMOSD, their families/carers and health care professionals (HCPs) will participate in interviews to gain perspectives and perceptions with regards to weight change, in order to develop a suitable intervention for implementation in the care pathway.

Design:

Participatory design with semi-structured interviews.

Objectives:

* Describe the factors affecting the management of these conditions, with regards to quality of life, health and wellbeing.
* Identify potential modifiable/non-modifiable factors that contribute to weight change in this population.
* Highlight and extract important concerns and themes, and explore the barriers and facilitators to implementing a lifestyle management system for this population within the care pathway.

Participants:

* 15 young people aged 10-25 with MS or NMOSD (Including MOG)
* 15 parents/carers.
* 15 health care practitioners from medical, nursing and AHP backgrounds with at least two years' experience in NMOSD and MS.
* N= 45.

Method:

Semi-structured interviews underpinned by a thematic analysis with patients, parents and clinicians. The questions will be focused around predetermined themes and factors, extracted from the previously performed scoping review and data audit, and involving nutrition, weight changes, overall health and quality of life. The team psychologist will co-develop questions related to behaviour, and The nutritionist and exercise specialist will co-develop in their respective fields. The PPI members will co-develop all interview formats and methods. There will be three different versions of the questions; one for patients, one for parents and one for clinicians. The interview questions will remain consistent throughout the study.

Procedure:

Interviews with parents, patients and HCP's will be performed virtually via video call, using the secured Google Hangouts platform. Invitations to join the link will be sent via email, and events will be made private.

The participants will have the option to participate while at home, or at one of the three research sites during one of their clinical appointment days. It is foreseen that patients and their parents will participate virtually from their home, however, should they need assistance or accommodation, this will be provided by one of our three research sites. In this case, the clinical nurse will assist with the virtual interview, when the patient is present at one of the hospitals for their bi-yearly day of clinical appointments. Clinicians will also be given the option to either participate virtually from home, or from one of the research sites. The interviewer will perform the interview from a private room at Oxford Brookes University. Parents will be interviewed on their own, whereas patients will be interviewed with their parent present- if under 16. Patients aged 16+ years may have their parents present should they wish, but the parent will be asked not to contribute. The estimated interview time is 45- 60 mins, subject to change during the development process. There will be a brief post interview questionnaire where the participants will be given the opportunity to mention anything they might not have been able to discuss in the interview. It will also allow for the research team to collect data with regards to the execution of the research and to consequently assess the chosen methods.

Analysis:

Interviews will be recorded using a secured Google Hangouts platform to provide accurate accounts of participant discussions and then transcribed verbatim and checked for accuracy. Only the audio component of the interview will be recorded, not the video component, in order to protect the privacy of participants. The design, conduct and dissemination of this research will be guided by the COREQ Checklist. Semi-structured interviews will be guided with an interview schedule and topic guide. Recordings will be transcribed by the third party transcription company: Rapid Transcriptions . The investigators will take a subtle realist position to allow the inclusion of a-priori knowledge and use an inductive thematic analysis. To report themes and patterns within the data. NVivo 12 for Windows will be used to assist with the organisation and retrieval of data. The design, conduct, and dissemination will be guided by the COREQ Checklist. The transcripts will be read by two of the team.

Considerations:

The investigators will use young people friendly age applicable materials and tools to facilitate conversations such as TALKING- MATs; a system in which the participant can use pictures or actions and answers in order to help facilitate their communication. A pre-interview questionnaire will be performed to inform the interviewer of patient status prior to starting. A traffic light system will also be introduced, to allow the patient to express their desire to stop the interview if they feel the need to.

Phase 2: Logic model of factors.

Objectives:

* To establish a list of factors that contribute to weight change in paediatric MS and NMOSD patients.
* To create a logic model of the problem and contributing factors.

Methods:

The research team will integrate the findings from the first three stages of the program of work including background foundation work (review, and audit) and the Phase 1 interviews (perspectives of patients, families and clinicians). A list of factors that contribute to weight changes in this population will be identified based on the extraction of data form the previously completed scoping review, data audit, and the interviews completed in the previous stage. In keeping with the Intervention Mapping methodology structuring this research project, a logic model will be created. These factors will be in the domains of environment, behaviour, clinical features and treatment.

Phase 3: Stakeholder Meetings.

Objectives:

* Obtain input from a stakeholder panel to decide measures, factors and outcomes
* Finalise the content and delivery protocols of the intervention.
* Co-design the program and context of use including delivery systems and content to sit within the care pathway.

Participants:

•N=12 (4 clinicians, 4 parent, 4 young people with MS or NMOSD)

Participants from Phase 1 and the research team will be invited to participate considering the same inclusion/exclusion criterion. Four parent and patients members will attend the meetings with our research team in person, while four our consulting clinicians will attend the meeting via video call through the Google Hangouts platform.

Methods:

The logic model created in Phase 2, which outlines all the identifiable factors that contribute to weight change will be presented to the panel of key stakeholders in co-production workshops. There will be two workshops in the form of meetings. These will be run on a virtual platform, via Google Hangouts, and ideas recorded using a virtual whiteboard. No audio or video recordings will be taken. Real-time Board inc (Miro) is compliant with GDPR and is registered and certified with the Cloud security alliance https://cloudsecurityalliance.org/star/registry/realtimeboard-inc/ for meeting industry standards.

Meeting 1 development: This meeting will review and identify outcomes in order to finalize content by bringing together evidence from the literature, clinical data and the perspectives of patients, families and clinicians. The investigators will use a modified nominal group approach following the steps: preparation of logistics/focus, silent idea generation, round-robin recording of ideas, serial discussion of ideas, preliminary consensus formation, discussion and final agreement of logic model, and intervention and evaluation plan and intervention. Provisional program outcomes and objectives will be established, and a logic model of change. The research team will then co-design the lifestyle weight management program by generating program themes, components, and delivery protocols.

Meeting 2 consensus: The program and its themes, components and protocols will then be presented to the panel during the second meeting. The same nominal group methodology will be used as in the first session. Feedback will be obtained regarding recruitment, participation, implementation and adherence in order to put forth the most appealing program for patients, parents, clinicians and researchers. Following the second meeting adjustments to the program will be made, so that it is ready for the feasibility stage.

STUDY SETTING Phase 1: Interviews.

This is a multi-centre study and will involve virtually interviewing patients, parents and clinicians at their homes, or at one of our three sites, listed below:

John Radcliffe Hospital, Oxford, UK. Great Ormond Street Hospital, London, UK. Evelina Hospital, London, UK. The decision to conduct interviews through these sites was made with the patient in mind, as the data collection will be integrated into the patients' bi-annual clinic in which they travel to the hospital(s) for the completion of several appointments. The interview will last approximately 45-60 minutes and will be in-cooperated into their appointment schedule for that day. Furthermore, as the patients regularly attend these hospitals, the research site will be familiar to them. The interviewee will be set up in a room located on one of the three aforementioned study sites, or at their home. This option has been added in order to accommodate for any participants that might not deem it safe enough to visit one of the three research sites during the current status of the COVID global pandemic. The decision to perform the interviews virtually was made following current COVID guidelines, in order to protect both interviewer and interviewee through the limitation of contact and consequently lowering of risk. The interviewer will be located in a private room at Oxford Brookes University. Recruitment will also occur at these three sites, and will be performed by the clinical nurse associated to the appropriate MS/NMOSD team at each site prior to the scheduled interview days.

Phase 3: Stakeholder Meetings This phase of the research will occur virtually via the same Google Hangouts platform as Phase 1. Participants will be asked to attend two stakeholder meetings occurring on two different days.

Sample identification and recruitment Phase 1: Interviews Potential eligible participants (young people and their parents) will be identified by the clinical nurse located at each of our three research sites (JR in Oxford, GOSH and Evelina in London) from their current list of patients. The role of the nurse will involve participant identification and eligibility checks. Once potential participants have been identified, the clinical nurse will mail out a patient information package (containing research team contact information) alongside their bi-annual appointment reminder. The potential participants will then have the option to opt into the study. Potential health care practitioners will be identified by our lead clinicians and clinical nurses, and will be contacted by the research nurse via email.

Phase 3: Stakeholder Meetings Participants (young people and parents) for phase 3 will be existing participants recruited from those who participated in Phase 1. During the consent procedure for phase 1, the participants will have the option to consent to being contacted by the research team regarding future research; those who consent will be recruited for phase 3. Health care professionals that are currently members of our advisory team will be included. No further recruitment will be necessary.

Consent Informed Consent The participant must sign and date the latest approved version of the Informed Consent form, before any study specific procedures occur.

Written and verbal versions of the Participant Information and Informed Consent will be presented to the participants detailing no less than: the exact nature of the trial; what it will involve for the participant; the implications and constraints of the protocol; the known side effects and any risks involved in taking part. It will be clearly stated that the participant is free to withdraw from the trial at any time for any reason without prejudice to future care, without affecting their legal rights and with no obligation to give the reason for withdrawal.

The participant will be allowed as much time as wished to consider the information, and the opportunity to question the Investigator, their GP or other independent parties to decide whether they will participate in the trial. Written Informed Consent will then be obtained by means of participant dated signature and dated signature of the person who presented and obtained the Informed Consent. Informed assent will be sought from any participant aged 10-15, as well as informed consent from their parent/guardian. There will be child friendly Participant Information Sheets catered for those aged 10-15, so as to assure their assent is well informed. The person who obtained the consent must be suitably qualified and experienced, and have been authorised to do so by the Chief/Principal Investigator. A copy of the signed Informed Consent will be given to the participant. The original signed form will be retained at the trial site. Outcomes will be analysed after recruitment of the last participant in the trial. Phase 1 of the study will close once the final participant has completed their interview. Informed consent for Phase 3 will commence after the completion of Phase 1, and the informed consent procedure will remain the same.

Withdrawal and loss to follow-up Parents/ guardians of participants, and the participants, have the right to withdraw consent/assent for participation in any aspect of this trial at any time. Routine medical care will not be affected at any time by declining to participate or withdrawing from the trial. The investigators will make every effort to reduce loss to follow-up. One primary contact within each centre will contact all participants and act as liaison with the assessor and therapy team. The primary contact person will obtain information about the participants' preferred method of contact (text, telephone, email, and letter) and trial researchers will contact them using this preferred method when possible. Contact details will be updated if applicable at each assessment. All appointments will be made at the research participant's convenience wherever possible. If an appointment is missed the investigators will try to rearrange this on one more occasions.

ELIGIBILITY:
Inclusion Criteria:

* Patients:
* Age 10-25 years
* Diagnosis of MS or NMOSD (including MOG) prior to 18 years
* Living in England or Wales
* Currently monitored by the JR in Oxford, or GOSH or Evelina in London
* With the capacity to assent/ consent Parents
* Parent of a young person with MS or NMOSD (including MOG)
* Child must have been diagnosed prior to the age of 18
* Living in England or Wales
* With the capacity to consent Clinicians
* Health care practitioner from medical, nursing and AHP backgrounds
* With at least two years' experience working in MS and NMSOD clinics (adult or paediatric).

Exclusion Criteria:

* Unable to give informed consent
* Unable to communicate or participate safely (as determined by themselves or their parents/carers)

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will see a total of 57 participants (some repeated) over the course of phase 1 and phase 3. Phase 1 will include a sample size of n=45: 15 young people, 15 parents and 15 clinicians. Phase 3 will include 4 parent, 4 patient, and 4 clinicians for a total of n=12.
  As these are rare conditions, with complicated diagnostic criteria, it is difficult to obtain exact national figures; however it is estimated that 200 young people across the UK have relapsing demyelinating syndromes (RDS). This figure includes MS and NMOSD cases, but also includes other such as CID, but only accounts for patients aged 18 and under. It is very difficult to provide an accurate number of patients aged 10-25 with MS or NMOSD who have been diagnosed prior to the age of 18. The three PIC sites associated with this study are part of the national MS and NMOSD services, and there is currently a combined total of 64 MS patients aged 10-18, and 73 NMOSD cases aged 10-18; for a total of n=137.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Lifestyle interviews: Themes and factors. | 6 months from start
  The interview phase of this research will output a list of factors reported by patients, parents and clinicians with regards to lifestyle change following their diagnosis. The investigators will measure the factors and themes most frequently identified by the interviewees and will assess themes through thematic analysis. Recruitment will also be assessed as well as overall participant experience.

CONTACTS AND LOCATIONS:
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No